CLINICAL TRIAL: NCT00006160
Title: African-American Diabetes Intervention Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: dahmsw (completed); DK48163
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Insulin-Dependent Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Behavioral: home based worker

SUMMARY:
A controlled trial to assess the potential benefit of a home based worker in improving control in African-American children with insulin dependent diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Insulin dependent diabetes mellitus

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States